CLINICAL TRIAL: NCT01737801
Title: Time to Perform Lung Function Test in Cystic Fibrosis After Chest Physiotherapy.
Brief Title: Time to Perform Lung Function Test in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Cecilia Rodriguez, Physiotherapist, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-CF-2
Record Dates: First submitted 2012-11-19; First posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Cystic Fibrosis
Keywords: Lung function; Physiotherapy
MeSH Terms: conditions — Cystic Fibrosis | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lung function test (Experimental): Lung function test
  Interventions: Procedure: Lung function test

INTERVENTIONS:
Procedure: Lung function test — Lung function test.
  Other Names: Lung function test.

SUMMARY:
Time to perform lung function test after chest physiotherapy in cystic fibrosis.

The investigators study FEV1(forced expiratory volume in one second) and FVC (forced vital capacity).

DETAILED DESCRIPTION:
The patients perform spirometry before, direct after, 30 minutes, 1 hour, 2 hours, and 3 hours after physiotherapist. The investigators want to study the FEV1 and FVC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cystic fibrosis

Exclusion Criteria:

* patients with cystic fibrosis who could not stay at the clinic for more than 4 hrs.

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-02; Primary Completion 2012-01 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Lung function test. FEV1 and FVC | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Rodriguez, Physio, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Stockholm, Stockholm County, Sweden